CLINICAL TRIAL: NCT03211377
Title: Non-interventional Study to Evaluate Chemotherapy for Potentially Resectable Locally Advanced Esophagogastric Junction Carcinoma
Brief Title: Chemotherapy for Potentially Resectable Locally Advanced Esophagogastric Junction Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anyang Tumor Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TOTMSEJ1701
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Esophagogastric Junction Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- neoadjuvant therapy group: Preoperation chemotherapy treatment for patients up to four cycles
- adjuvant therapy: Postoperation chemotherapy treatment for patients up to six cycles
- Perioperative therapy: Preoperation chemotherapy treatment for patients up to four cycles and postoperation chemotherapy up to six cycles

SUMMARY:
This is a non-interventional study to observe the safety and efficiency of chemotherapy for potentially resectable locally advanced esophagogastric junction

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological proved locally advanced esophagogastric junction cancer
* ECOG performance status ≦2
* Stage IIa-IIIc
* No distant metastasis (M0)
* Sign in Informed Consent Form

Exclusion Criteria:

* History of hypersensitivity to fluoropyrimidines, Tegafur，Gimeracil and Oteracil Potassium Capsules , capecitabine, oxaliplatin or the ingredients of this product
* Pregnancy or lactation women,
* Inadequate hematopoietic function： WBC≦3,500/mm3; ANC≦1,500/mm3; Platelet≦80,000/mm3
* Inadequate organ function which is defined as below:

Total bilirubin >2 pper limit of normal range (ULN); ALT / AST > 2.5 upper limit of normal range (ULN); serum creatinine > 1.5 mg/dL, and Ccr > 60 ml/min (estimated by Cockcroft-Gault formulation);

* Symptomatic peripheral neuropathy
* Receiving a concomitant treatment with other fluoropyrimidines
* Fluoropyrimidines (DPD) congenital absence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study patients had to be at least 18 years old with histologically or cytologically confirmed locally advanced esophagogastric junction cancer
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-03-29 (Estimated); Study Completion 2021-04-29 (Estimated)

PRIMARY OUTCOMES:
disease free survival(DFS) | up to 3 years
  time from surgery to disease recurrence or death

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  time to death
Adverse events(AE) | through study completion, up to 1 year
  Investigators graded all adverse events and toxic effects according to the National Cancer Institute's Common Toxicity Criteria, version 4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of science and education, Anyang, Henan, China